CLINICAL TRIAL: NCT02599402
Title: Clinical Trial of Nivolumab (BMS-936558) Combined With Ipilimumab Followed by Nivolumab Monotherapy as First-Line Therapy of Subjects With Histologically Confirmed Stage III (Unresectable) or Stage IV Melanoma CheckMate 401: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 401
Brief Title: Nivolumab Combined With Ipilimumab Followed by Nivolumab Monotherapy as First-Line Treatment for Patients With Advanced Melanoma
Acronym: CheckMate 401
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-401; 2015-001274-17 (EudraCT Number)
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combination therapy: Nivolumab + Ipilimumab (Experimental): Nivolumab + Ipilimumab specified dose on specified days
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Monotherapy: Nivolumab (Experimental): Nivolumab specified dose on specified days
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
Drug: Ipilimumab
  Arms: Combination therapy: Nivolumab + Ipilimumab

SUMMARY:
The purpose of this study is to determine the effects of combination treatment of Nivolumab with Ipilimumab followed by Nivolumab monotherapy in patients with previously untreated advanced Melanoma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Potential subjects must have advanced Melanoma (stage III or IV as confirmed by biopsy) with spread to other sites in the body and unable to be removed by surgery.
* Potential subjects must be newly diagnosed with advanced melanoma and received no treatment for the advanced disease.

NOTE: Prior adjuvant or neoadjuvant melanoma therapy (including anti-CTLA-4, anti-PD-1, anti-PD-L1, anti-PD-L2, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways, such as anti-CD-137) is permitted if the therapy was used in the adjuvant or neoadjuvant setting but not in the metastatic setting. These drugs must be discontinued 6 months prior to study entry and the side effects related to the prior therapy resolved.

* Potential subjects (with disease spread to brain) who previously received primary treatment are permitted if there was no evidence of disease as confirmed by the MRI (at least 2 weeks after the primary treatment is complete and with in 6 weeks of the first dose of the study drug). Potential subjects must not have received intravenous steroid treatment (>10 mg/day) intravenously for at least 2 weeks prior to study drug administration.

Exclusion Criteria:

* Leptomenigeal metastases
* Subjects with autoimmune disease. Subjects with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* All side effects from previous primary treatments other than alopecia, fatigue, or peripheral neuropathy must have resolved to Grade 1 or baseline before administration of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2015-12-20 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (103):
- Australia (16):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Coffs Harbour, New South Wales
  - Local Institution, Gateshead, New South Wales
  - Local Institution, North Sydney, New South Wales
  - Local Institution, Tiwi, Northern Territory
  - Local Institution, Brisbane, Queensland
  - Local Institution, Cairns, Queensland
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Southport, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Hobart, Tasmania
  - Local Institution, Melbourne, Victoria
  - Local Institution, Murdoch, Western Australia
  - Local Institution, Nedlands, Western Australia
- Austria (4):
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Salzburg
  - Local Institution, Vienna
- Local Institution, Brussels, Belgium
- Finland (4):
  - Local Institution, Helsinki
  - Local Institution, Oulu
  - Local Institution, Tampere
  - Local Institution, Turku
- France (19):
  - Local Institution, Angers
  - Local Institution, Bordeaux
  - Local Institution, Boulogne-Billancourt
  - Local Institution, Clermont-Ferrand
  - Local Institution, Dijon
  - Local Institution, Grenoble
  - Local Institution, Le Mans
  - Local Institution, Lille
  - Local Institution, Marseille
  - Local Institution, Montpellier
  - Local Institution, Nantes
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pierre Benite Cedax
  - Local Institution, Rennes
  - Local Institution, Rouen
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
  - Local Institution, Villejuif
- Germany (17):
  - Local Institution, Mainz, Rhineland-palladium
  - Local Institution, Berlin
  - Local Institution, Dresden
  - Local Institution, Erfurt
  - Local Institution, Erlangen
  - Local Institution, Frankfurt
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Göttingen
  - Local Institution, Hanover
  - Local Institution, Kiel
  - Local Institution, Leipzig
  - Local Institution, Ludwigshafen
  - Local Institution, Lübeck
  - Local Institution, Mannheim
  - Local Institution, Regensburg
  - Local Institution, Schwerin
  - Local Institution, Stade
- Ireland (3):
  - Local Institution, Cork
  - Local Institution, Dublin
  - Local Institution, Galway
- Italy (12):
  - Local Institution, Bari
  - Local Institution, Bergamo
  - Local Institution, Genova
  - Local Institution, Meldola
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Siena
  - Local Institution, Terni
  - Local Institution, Torino
- Norway (2):
  - Local Institution, Oslo
  - Local Institution, Stavanger
- Sweden (8):
  - Local Institution, Eskilstuna
  - Local Institution, Gävle
  - Local Institution, Karlskrona
  - Local Institution, Linköping
  - Local Institution, Stockholm
  - Local Institution, Sundsvall
  - Local Institution, Vaxjo
  - Local Institution, Västerås
- Switzerland (2):
  - Local Institution, Basel
  - Local Institution, Lausanne
- United Kingdom (15):
  - Local Institution, London, Greater London
  - Local Institution, Newcastle upon Tyne, Tyne and Wear
  - Local Institution, Cambridge
  - Local Institution, Cottingham
  - Local Institution, Glasgow
  - Local Institution, Headington
  - Local Institution, London
  - Local Institution, Manchester
  - Mount Vernon Hospital, Northwood
  - Local Institution, Nottingham
  - Local Institution, Preston
  - Local Institution, Sheffield
  - Local Institution, Southampton
  - Local Institution, Swansea
  - Local Institution, Truro

REFERENCES:
- [Derived] Dummer R, Corrie P, Gutzmer R, Meniawy TM, Del Vecchio M, Lebbe C, Guida M, Dutriaux C, Dreno B, Meyer N, Ferrucci PF, Dalle S, Khattak MA, Grob JJ, Briscoe K, Larkin J, Mansard S, Lesimple T, Guidoboni M, Sabatini S, Richtig E, Herbst R, Lobo M, Askelson M, Ascierto PA, Maio M. First-Line, Fixed-Duration Nivolumab Plus Ipilimumab Followed by Nivolumab in Clinically Diverse Patient Populations With Unresectable Stage III or IV Melanoma: CheckMate 401. J Clin Oncol. 2023 Aug 10;41(23):3917-3929. doi: 10.1200/JCO.22.02199. Epub 2023 Jun 12. PMID 37307514
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 533 participants treated
Groups:
- Nivolumab + Ipilimumab Total: Part 1: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240 mg) IV Q2W up to 21 months
Period: Overall Study
Arm/Group | Nivolumab + Ipilimumab Total
Started | 533
Completed | 0
Not Completed | 533
Not completed — Disease progression | 153
Not completed — Study drug toxicity | 201
Not completed — Death | 26
Not completed — Adverse Event unrelated to study drug | 23
Not completed — Participant request to discontinue study treatment | 13
Not completed — Participant withdrew consent | 5
Not completed — Lost to Follow-up | 1
Not completed — Maximum Clinical Benefit | 7
Not completed — Poor/non-compliance | 1
Not completed — Pregnancy | 1
Not completed — Participant no longer met study criteria | 7
Not completed — Other Reasons | 95

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab + Ipilimumab Total
Number analyzed (Participants) | 533
Age, Continuous [Median (Standard Deviation); unit: Years] | 59.0 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217
  Male | 316
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 515
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 521
  More than one race | 0
  Unknown or Not Reported | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Participants With High-Grade (CTCAE v4.0 Grade 3-5) Treatment-Related Select Adverse Events
Description: Incidence of participants with high-grade (CTCAE v4.0 grade 3-5) treatment-related, select adverse events of potentially immune-mediated etiology including pulmonary, gastrointestinal, skin, renal, hepatic, endocrine, infusion-related, or hypersensitivity
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups
Measure: Count of Participants; unit: Participants
Groups:
- Nivolumab + Ipilimumab Total: Part 1: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
- Nivolumab + Ipilimumab ECOG PS0-1: Part 1: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1 subgroup
- Nivolumab + Ipilimumab ECOG PS2: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2 subgroup
- Nivolumab + Ipilimumab Brain Metastasis: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Brain Metastasis subgroup
- Nivolumab + Ipilimumab Mucosal: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Disease Subtype subgroup Mucosal
- Nivolumab + Ipilimumab Ocular/Uveal: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Disease Subtype subgroup Ocular/Uveal
- Nivolumab + Ipilimumab Cutaneous: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Disease Subtype subgroup Cutaneous
- Nivolumab + Ipilimumab Acral: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Disease Subtype subgroup Acral
- Nivolumab + Ipilimumab Other: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses up to 3 months
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W up to 21 months
  Participants were grouped in to Disease Subtype subgroup Other
Arm/Group | Nivolumab + Ipilimumab Total | Nivolumab + Ipilimumab ECOG PS0-1 | Nivolumab + Ipilimumab ECOG PS2 | Nivolumab + Ipilimumab Brain Metastasis | Nivolumab + Ipilimumab Mucosal | Nivolumab + Ipilimumab Ocular/Uveal | Nivolumab + Ipilimumab Cutaneous | Nivolumab + Ipilimumab Acral | Nivolumab + Ipilimumab Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Participants
  Pulmonary: Grade 3-4 | 7 | 7 | 0 | 0 | 0 | 1 | 6 | 0 | 0
  Pulmonary: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal: Grade 3-4 | 83 | 79 | 4 | 5 | 5 | 9 | 57 | 1 | 11
  Gastrointestinal: Grade 5 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Skin: Grade 3-4 | 35 | 31 | 4 | 1 | 3 | 7 | 20 | 1 | 4
  Skin: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Renal: Grade 3-4 | 10 | 9 | 1 | 1 | 0 | 1 | 8 | 0 | 1
  Renal: Grade 5 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hepatic: Grade 3-4 | 82 | 75 | 7 | 6 | 2 | 17 | 56 | 1 | 6
  Hepatic: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Endocrine: Grade 3-4 | 58 | 58 | 0 | 5 | 2 | 6 | 43 | 1 | 6
  Endocrine: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypersensitivity/Infusion Reaction: Grade 3-4 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypersensitivity/Infusion Reaction: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Incidence of Participants With All High-Grade (Grades 3-5) Select Adverse Events
Description: Incidence of participants with high-grade (grade 3-5) select adverse events including pulmonary, gastrointestinal, skin, renal, hepatic, infusion-related, or hypersensitivity
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups
Measure: Count of Participants; unit: Participants
Groups:
- Total: Part 1: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W
- ECOG PS0-1: Part 1: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W
- ECOG PS2; Brain Metastasis; Mucosal; Ocular/Uveal; Cutaneous; Acral; Other: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Participants
  Pulmonary: Grade 3-4 | 8 | 8 | 0 | 0 | 0 | 1 | 7 | 0 | 0
  Gastrointestinal: Grade 3-4 | 87 | 83 | 4 | 5 | 5 | 9 | 61 | 1 | 11
  Gastrointestinal: Grade 5 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Skin: Grade 3-4 | 39 | 35 | 4 | 1 | 3 | 8 | 22 | 1 | 5
  Renal: Grade 3-4 | 13 | 12 | 1 | 1 | 0 | 1 | 10 | 1 | 1
  Renal: Grade 5 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hepatic: Grade 3-4 | 101 | 93 | 8 | 11 | 4 | 21 | 67 | 1 | 8
  Hepatic: Grade 5 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypersensitivity/Infusion Reaction: Grade 3-4 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1

3. Secondary Outcome: Median Time to Onset (Grades 3-4) of Select Adverse Events
Description: Median time to onset (grades 3-4) of select adverse events including pulmonary, gastrointestinal, skin, renal, hepatic, endocrine, infusion-related, or hypersensitivity
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups with at least one select adverse event from the category
Measure: Median (Full Range); unit: Days
Groups:
- Total; ECOG PS0-1: Part 1: Nivolumab 1 mg/kg IV + Ipilimumab 3 mg/kg IV Q3W x 4 doses
  Then
  Part 2: Nivolumab (3mg/kg or 240mg) IV Q2W
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Days
  Pulmonary: number analyzed (Participants) | 8 | 8 | 0 | 0 | 0 | 1 | 7 | 0 | 0
  Pulmonary | 51.5 [12 to 783] | 51.5 [12 to 783] |  |  |  | 51.0 [51 to 51] | 52.0 [12 to 783] |  |
  Gastrointestinal: number analyzed (Participants) | 88 | 84 | 4 | 42 | 6 | 9 | 61 | 10 | 11
  Gastrointestinal | 49.0 [7 to 582] | 49.0 [7 to 582] | 61.0 [8 to 91] | 83.0 [35 to 543] | 42.5 [27 to 543] | 39.0 [20 to 95] | 49.0 [7 to 582] | 7.0 [7 to 7] | 79.0 [8 to 281]
  Skin: number analyzed (Participants) | 39 | 35 | 4 | 1 | 3 | 8 | 22 | 1 | 5
  Skin | 32.0 [4 to 670] | 35.0 [4 to 404] | 17.5 [7 to 670] | 14.0 [14 to 14] | 48.0 [8 to 69] | 36.5 [14 to 127] | 17.5 [4 to 670] | 89.0 [89 to 89] | 100.0 [10 to 338]
  Renal: number analyzed (Participants) | 14 | 13 | 1 | 1 | 0 | 1 | 11 | 1 | 1
  Renal | 52.5 [6 to 540] | 43.0 [6 to 223] | 540.0 [540 to 540] | 106.0 [106 to 106] |  | 23.0 [23 to 23] | 106.0 [14 to 540] | 16.0 [16 to 16] | 6.0 [6 to 6]
  Hepatic: number analyzed (Participants) | 102 | 94 | 8 | 11 | 4 | 22 | 67 | 1 | 8
  Hepatic | 63.0 [5 to 724] | 63.0 [5 to 724] | 63.0 [13 to 83] | 64.0 [41 to 724] | 139.0 [22 to 475] | 64.0 [16 to 111] | 62.0 [5 to 588] | 101.0 [101 to 101] | 80.0 [8 to 724]
  Endocrine: number analyzed (Participants) | 59 | 59 | 0 | 5 | 2 | 6 | 44 | 1 | 6
  Endocrine | 75.0 [7 to 369] | 75.0 [7 to 369] |  | 67.0 [25 to 130] | 153.0 [102 to 204] | 70.0 [26 to 98] | 71.5 [7 to 369] | 114.0 [114 to 114] | 39.5 [16 to 115]
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hypersensitivity/Infusion Reaction | 291.5 [22 to 561] | 291.5 [22 to 561] |  |  |  |  | 22.0 [22 to 22] |  | 561.0 [561 to 561]

4. Secondary Outcome: Median Time to Resolution (Grades 3-4) of Select Adverse Events
Description: Median time to resolution (Grades 3-4) of select adverse events including pulmonary, gastrointestinal, skin, renal, hepatic, endocrine, infusion-related, or hypersensitivity
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Days
  Pulmonary: number analyzed (Participants) | 8 | 8 | 0 | 0 | 0 | 1 | 7 | 0 | 0
  Pulmonary | 19.0 [5 to 64] | 19.0 [5 to 64] |  |  |  | 6.0 [6 to 6] | 30.0 [5 to 64] |  |
  Gastrointestinal: number analyzed (Participants) | 88 | 84 | 4 | 5 | 6 | 9 | 61 | 1 | 11
  Gastrointestinal | 22.0 [2 to 684] | 22.0 [2 to 684] | NA [8 to 437] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 107.5 [18 to 666] | 25.0 [6 to 437] | 14.0 [6 to 183] | 23.0 [2 to 684] | 5.0 [5 to 5] | 12.0 [4 to 214]
  Skin: number analyzed (Participants) | 39 | 35 | 4 | 1 | 3 | 8 | 22 | 1 | 5
  Skin | 24.0 [4 to 690] | 24.0 [4 to 690] | 20.0 [10 to 186] | 67.0 [67 to 67] | 8.0 [5 to 44] | 17.5 [4 to 690] | 24.0 [8 to 455] | 15.0 [15 to 15] | 28.0 [4 to 287]
  Renal: number analyzed (Participants) | 14 | 13 | 1 | 1 | 0 | 1 | 11 | 1 | 1
  Renal | 19.0 [3 to 66] | 23.0 [3 to 66] | 11.0 [11 to 11] | 7.0 [7 to 7] |  | 23.0 [23 to 23] | 11.0 [3 to 60] | NA [20 to 20] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 66.0 [66 to 66]
  Hepatic: number analyzed (Participants) | 102 | 94 | 8 | 11 | 4 | 22 | 67 | 1 | 8
  Hepatic | 42.0 [1 to 889] | 38.0 [1 to 889] | 67.0 [3 to 225] | 17.5 [2 to 285] | 126.0 [1 to 625] | 55.0 [1 to 612] | 30.0 [2 to 889] | 29.0 [29 to 29] | 117.0 [15 to 285]
  Endocrine: number analyzed (Participants) | 59 | 59 | 0 | 5 | 2 | 6 | 44 | 1 | 6
  Endocrine | NA [2 to 1223] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [3 to 1019] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. |  | NA [4 to 950] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [5 to 931] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [3 to 670] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [4 to 1019] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [514 to 514] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [4 to 627] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits.
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hypersensitivity/Infusion Reaction | 4.5 [2 to 7] | 4.5 [2 to 7] |  |  |  |  | 2.0 [2 to 2] |  | 7.0 [7 to 7]

5. Secondary Outcome: Time to Resolution of an Adverse Event (AE)
Description: Resolution of an adverse event (AE) is defined as a participant experiencing complete resolution or improvement to the baseline of any grade AE including pulmonary, gastrointestinal, skin, renal, hepatic, endocrine, infusion-related, or hypersensitivity
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Days
  Pulmonary: number analyzed (Participants) | 28 | 26 | 2 | 2 | 2 | 3 | 21 | 0 | 2
  Pulmonary | 35.0 [6 to 738] | 43.0 [6 to 738] | 7.5 [7 to 8] | NA [55 to 302] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [7 to 371] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 19.0 [6 to 62] | 43.0 [7 to 738] |  | NA [24 to 302] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits.
  Gastrointestinal: number analyzed (Participants) | 252 | 236 | 16 | 14 | 13 | 31 | 175 | 6 | 27
  Gastrointestinal | 18.0 [1 to 1016] | 18.0 [1 to 1016] | 12.0 [1 to 468] | 36.0 [1 to 720] | 14.0 [1 to 527] | 14.0 [1 to 183] | 19.0 [1 to 1016] | 5.0 [1 to 22] | 36.0 [2 to 645]
  Skin: number analyzed (Participants) | 319 | 296 | 23 | 23 | 17 | 34 | 228 | 8 | 32
  Skin | 89.0 [1 to 1175] | 88.0 [1 to 1175] | NA [5 to 1002] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 257.0 [1 to 1011] | 84.0 [5 to 1055] | 33.5 [4 to 775] | 102.0 [1 to 1175] | 46.0 [15 to 625] | 59.5 [2 to 952]
  Renal: number analyzed (Participants) | 43 | 42 | 1 | 4 | 2 | 2 | 34 | 1 | 4
  Renal | 56.0 [2 to 904] | 56.0 [2 to 904] | 11.0 [11 to 11] | 5.5 [2 to 100] | 9.5 [4 to 15] | 27.5 [23 to 32] | 56.0 [2 to 904] | NA [20 to 20] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [66 to 603] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits.
  Hepatic: number analyzed (Participants) | 185 | 173 | 12 | 16 | 7 | 35 | 128 | 2 | 13
  Hepatic | 44.0 [1 to 1008] | 43.0 [1 to 1008] | 80.5 [3 to 225] | 20.5 [3 to 1008] | 97.0 [1 to 650] | 34.0 [1 to 612] | 37.0 [3 to 912] | 129.0 [31 to 129] | 29.0 [8 to 1008]
  Endocrine: number analyzed (Participants) | 242 | 231 | 11 | 20 | 15 | 29 | 166 | 5 | 27
  Endocrine | NA [2 to 1223] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [2 to 1223] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [76 to 917] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [4 to 950] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [5 to 1139] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [2 to 759] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [4 to 1223] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [40 to 938] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [6 to 1060] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits.
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 8 | 7 | 1 | 0 | 0 | 0 | 5 | 0 | 3
  Hypersensitivity/Infusion Reaction | 1.0 [1 to 7] | 1.0 [1 to 7] | 1.0 [1 to 1] |  |  |  | 1.0 [1 to 7] |  | 1.0 [1 to 7]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined from the time of first dosing date to the date of death. A participant who has not died will be censored at the last known date alive
Time Frame: Up to approximately 37 months
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Months | NA [33.91 to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [34.76 to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 11.01 [7.23 to NA] — Insufficient data due to insufficient participant follow up. | NA [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 12.55 [3.78 to 33.91] | 15.21 [10.41 to 21.42] | NA [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 20.83 [1.15 to NA] — Insufficient data due to insufficient participant follow up. | 34.76 [16.69 to NA] — Insufficient data due to insufficient participant follow up.

7. Secondary Outcome: Incidence of Participants With Adverse Events
Description: The assessment of safety is measured by the incidence of participants who experienced any grade of adverse events (AEs), treatment-related AEs, serious adverse events (SAEs), and deaths
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Participants
  Adverse Events (AEs) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
  Treatment-Related AEs | 484 | 444 | 40 | 33 | 26 | 61 | 332 | 8 | 35
  Serious Adverse Events (SAEs) | 356 | 324 | 31 | 31 | 26 | 40 | 238 | 9 | 43
  Deaths | 199 | 169 | 29 | 13 | 20 | 41 | 107 | 6 | 25

8. Secondary Outcome: Incidence of Participants With Select Adverse Events
Description: The assessment of safety is measured by the incidence of participants who experienced any grade of select adverse events including pulmonary, gastrointestinal, skin, renal, hepatic, endocrine, infusion-related, or hypersensitivity
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Participants
  Pulmonary | 28 | 26 | 2 | 2 | 2 | 3 | 21 | 0 | 2
  Gastrointestinal | 252 | 236 | 16 | 14 | 13 | 31 | 175 | 6 | 27
  Skin | 319 | 296 | 23 | 23 | 17 | 34 | 228 | 8 | 32
  Renal | 43 | 42 | 1 | 4 | 2 | 2 | 34 | 1 | 4
  Hepatic | 185 | 173 | 12 | 16 | 7 | 35 | 128 | 2 | 13
  Endocrine | 242 | 231 | 11 | 20 | 15 | 29 | 166 | 5 | 27
  Hypersensitivity/Infusion Reaction | 8 | 7 | 1 | 0 | 0 | 0 | 5 | 0 | 3

9. Secondary Outcome: Incidence of Participants With Laboratory Abnormalities - Liver
Description: Safety assessment is measured by the incidence of participants who experienced a liver laboratory abnormality in Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Upper Limit of Normal (ULN)
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Participants
  ALT OR AST > 3XULN: number analyzed (Participants) | 490 | 442 | 48 | 37 | 29 | 56 | 338 | 10 | 57
  ALT OR AST > 3XULN | 113 | 106 | 7 | 11 | 7 | 21 | 72 | 2 | 11
  ALT OR AST > 5XULN: number analyzed (Participants) | 490 | 442 | 48 | 37 | 29 | 56 | 338 | 10 | 57
  ALT OR AST > 5XULN | 75 | 69 | 6 | 4 | 5 | 13 | 48 | 1 | 8
  ALT OR AST > 10XULN: number analyzed (Participants) | 490 | 442 | 48 | 37 | 29 | 56 | 338 | 10 | 57
  ALT OR AST > 10XULN | 30 | 27 | 3 | 0 | 2 | 4 | 22 | 0 | 2
  ALT OR AST > 20XULN: number analyzed (Participants) | 490 | 442 | 48 | 37 | 29 | 56 | 338 | 10 | 57
  ALT OR AST > 20XULN | 12 | 11 | 1 | 0 | 1 | 2 | 7 | 0 | 2
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 490 | 442 | 48 | 37 | 29 | 56 | 338 | 10 | 57
  TOTAL BILIRUBIN > 2XULN | 12 | 12 | 0 | 1 | 0 | 3 | 8 | 0 | 1
  CONCURRENT ALT OR AST ELEVATION > 3XULN; TOTAL BILIRUBIN > 2XULN IN 1 DAY: number analyzed (Participants) | 490 | 442 | 48 | 37 | 29 | 56 | 338 | 10 | 57
  CONCURRENT ALT OR AST ELEVATION > 3XULN; TOTAL BILIRUBIN > 2XULN IN 1 DAY | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  CONCURRENT ALT OR AST ELEVATION > 3XULN; TOTAL BILIRUBIN > 2XULN IN 30 DAYS: number analyzed (Participants) | 490 | 442 | 48 | 37 | 29 | 56 | 338 | 10 | 57
  CONCURRENT ALT OR AST ELEVATION > 3XULN; TOTAL BILIRUBIN > 2XULN IN 30 DAYS | 4 | 4 | 0 | 0 | 0 | 0 | 4 | 0 | 0

10. Secondary Outcome: Incidence of Participants With Laboratory Abnormalities - Thyroid
Description: Safety assessment is measured by the incidence of participants who experienced a thyroid laboratory abnormality in Free T3 (FT3), Free T4 (FT4), Lower Limit of Normal (LLN)
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups with at least one on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 449 | 410 | 39 | 35 | 26 | 49 | 313 | 10 | 51
Participants
  TSH > ULN | 130 | 123 | 7 | 12 | 8 | 12 | 91 | 4 | 15
  TSH > ULN WITH TSH <= ULN AT BASELINE | 113 | 108 | 5 | 11 | 6 | 10 | 79 | 3 | 15
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 80 | 76 | 4 | 8 | 5 | 6 | 55 | 2 | 12
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 37 | 35 | 2 | 3 | 1 | 4 | 27 | 2 | 3
  TSH > ULN WITH FT3/FT4 TEST MISSING | 26 | 25 | 1 | 2 | 2 | 2 | 21 | 0 | 1
  TSH < LLN | 178 | 169 | 9 | 14 | 11 | 23 | 124 | 4 | 16
  TSH <LLN WITH TSH >= LLN AT BASELINE | 168 | 159 | 9 | 14 | 11 | 21 | 116 | 4 | 16
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 101 | 98 | 3 | 7 | 8 | 12 | 72 | 2 | 7
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 59 | 53 | 6 | 5 | 3 | 8 | 40 | 1 | 7
  TSH < LLN WITH FT3/FT4 TEST MISSING | 26 | 25 | 1 | 2 | 0 | 4 | 19 | 1 | 2

11. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants with a best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of all treated participants
Time Frame: Up to approximately 37 months
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Percentage of participants | 44.5 [40.2 to 48.8] | 46.1 [41.6 to 50.7] | 30.9 [19.1 to 44.8] | 52.4 [36.4 to 68.0] | 43.8 [26.4 to 62.3] | 9.4 [3.5 to 19.3] | 51.2 [46.0 to 56.5] | 30.0 [6.7 to 65.2] | 43.5 [31.0 to 56.7]

12. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival per investigator assessment is defined as radiological evidence of progression, significant clinical symptomatic progression, or the need to introduce a non-study drug therapy.
Time Frame: Up to approximately 37 months
Population: All treated participants and ECOG, Brain Metastasis, and Disease Subtype subgroups
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total | ECOG PS0-1 | ECOG PS2 | Brain Metastasis | Mucosal | Ocular/Uveal | Cutaneous | Acral | Other
Number analyzed (Participants) | 533 | 477 | 55 | 42 | 32 | 64 | 365 | 10 | 62
Months | 4.96 [3.45 to 6.77] | 5.45 [3.78 to 7.69] | 2.46 [1.77 to 3.75] | 3.35 [1.81 to NA] — Insufficient data due to insufficient participant follow up. | 2.94 [2.53 to 8.74] | 2.83 [2.73 to 4.63] | 6.77 [4.67 to 10.45] | 2.56 [1.15 to 8.48] | 5.22 [2.76 to 27.27]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after last dose (up to approximately 37 months)
Arm/Group | Nivolumab + Ipilimumab Total | Nivolumab + Ipilimumab ECOG PS0-1 | Nivolumab + Ipilimumab ECOG PS2 | Nivolumab + Ipilimumab Brain Metastasis | Nivolumab + Ipilimumab Mucosal | Nivolumab + Ipilimumab Ocular/Uveal | Nivolumab + Ipilimumab Cutaneous | Nivolumab + Ipilimumab Acral | Nivolumab + Ipilimumab Other
All-Cause Mortality (participants affected / at risk) | 199/533 | 169/477 | 29/55 | 13/42 | 20/32 | 41/64 | 107/365 | 6/10 | 25/62
Serious Adverse Events (participants affected / at risk) | 356/533 | 324/477 | 31/55 | 31/42 | 26/32 | 40/64 | 238/365 | 9/10 | 43/62
Other Adverse Events (participants affected / at risk) | 503/533 | 453/477 | 49/55 | 37/42 | 28/32 | 61/64 | 347/365 | 10/10 | 57/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab Total (N=533) | Nivolumab + Ipilimumab ECOG PS0-1 (N=477) | Nivolumab + Ipilimumab ECOG PS2 (N=55) | Nivolumab + Ipilimumab Brain Metastasis (N=42) | Nivolumab + Ipilimumab Mucosal (N=32) | Nivolumab + Ipilimumab Ocular/Uveal (N=64) | Nivolumab + Ipilimumab Cutaneous (N=365) | Nivolumab + Ipilimumab Acral (N=10) | Nivolumab + Ipilimumab Other (N=62)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 3 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myocarditis (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 6 | 6 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 8 | 8 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Hypophysitis (Endocrine disorders) | 23 | 23 | 0 | 1 | 1 | 5 | 14 | 0 | 3
Hypopituitarism (Endocrine disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Immune-mediated hyperthyroidism (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 6 | 6 | 0 | 2 | 0 | 0 | 6 | 0 | 0
Primary adrenal insufficiency (Endocrine disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thyroiditis acute (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune uveitis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 12 | 11 | 1 | 1 | 1 | 1 | 6 | 1 | 3
Chronic gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 43 | 41 | 2 | 1 | 3 | 2 | 32 | 0 | 6
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 36 | 34 | 2 | 2 | 1 | 5 | 29 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 9 | 9 | 0 | 0 | 0 | 0 | 8 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Pancreatic failure (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Asthenia (General disorders) | 3 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthermia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polyserositis (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 14 | 14 | 0 | 1 | 1 | 2 | 10 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 15 | 14 | 1 | 1 | 0 | 2 | 12 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 4 | 4 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 3 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 8 | 7 | 1 | 0 | 3 | 1 | 3 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 3 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 15 | 15 | 0 | 2 | 0 | 3 | 9 | 0 | 3
Anaphylactic shock (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alveolar osteitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Bronchitis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 4 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 4 | 4 | 0 | 1 | 0 | 1 | 3 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumococcal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 4 | 0 | 1 | 0 | 2 | 2 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyoderma (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 6 | 5 | 1 | 1 | 0 | 0 | 5 | 1 | 0
Septic arthritis streptococcal (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Wound infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 6 | 0 | 0 | 1 | 2 | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical condition abnormal (Investigations) | 5 | 4 | 1 | 0 | 1 | 0 | 3 | 1 | 0
Liver function test increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 4 | 4 | 0 | 0 | 0 | 0 | 4 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 6 | 0 | 0 | 1 | 0 | 5 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 3 | 3 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 71 | 57 | 14 | 13 | 8 | 9 | 42 | 2 | 10
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune neuropathy (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Autonomic neuropathy (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Cubital tunnel syndrome (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 7 | 1 | 1 | 1 | 0 | 7 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 10 | 10 | 0 | 2 | 1 | 1 | 7 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Immune-mediated renal disorder (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 1 | 1 | 0 | 0 | 6 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0 | 1 | 0 | 1 | 4 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 0 | 0 | 0 | 1 | 7 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 1 | 1 | 0 | 3 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vein collapse (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab Total (N=533) | Nivolumab + Ipilimumab ECOG PS0-1 (N=477) | Nivolumab + Ipilimumab ECOG PS2 (N=55) | Nivolumab + Ipilimumab Brain Metastasis (N=42) | Nivolumab + Ipilimumab Mucosal (N=32) | Nivolumab + Ipilimumab Ocular/Uveal (N=64) | Nivolumab + Ipilimumab Cutaneous (N=365) | Nivolumab + Ipilimumab Acral (N=10) | Nivolumab + Ipilimumab Other (N=62)
Anaemia (Blood and lymphatic system disorders) | 57 | 50 | 7 | 2 | 2 | 6 | 35 | 3 | 11
Hyperthyroidism (Endocrine disorders) | 98 | 96 | 2 | 7 | 7 | 14 | 69 | 0 | 8
Hypophysitis (Endocrine disorders) | 30 | 27 | 3 | 3 | 1 | 1 | 25 | 0 | 3
Hypothyroidism (Endocrine disorders) | 110 | 104 | 6 | 8 | 9 | 10 | 73 | 2 | 16
Abdominal pain (Gastrointestinal disorders) | 73 | 71 | 2 | 2 | 3 | 8 | 52 | 2 | 8
Abdominal pain upper (Gastrointestinal disorders) | 36 | 33 | 3 | 3 | 3 | 8 | 22 | 2 | 1
Constipation (Gastrointestinal disorders) | 83 | 77 | 6 | 12 | 7 | 6 | 61 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 224 | 209 | 15 | 13 | 13 | 27 | 154 | 5 | 25
Dry mouth (Gastrointestinal disorders) | 51 | 50 | 1 | 2 | 2 | 5 | 37 | 1 | 6
Nausea (Gastrointestinal disorders) | 156 | 144 | 11 | 10 | 8 | 24 | 105 | 5 | 14
Vomiting (Gastrointestinal disorders) | 82 | 75 | 7 | 9 | 5 | 6 | 60 | 2 | 9
Asthenia (General disorders) | 96 | 82 | 14 | 8 | 5 | 11 | 63 | 2 | 15
Chills (General disorders) | 27 | 26 | 1 | 2 | 4 | 2 | 18 | 0 | 3
Fatigue (General disorders) | 178 | 173 | 5 | 12 | 9 | 18 | 129 | 1 | 21
Influenza like illness (General disorders) | 41 | 41 | 0 | 1 | 3 | 3 | 31 | 1 | 3
Oedema peripheral (General disorders) | 34 | 31 | 3 | 3 | 4 | 5 | 18 | 2 | 5
Pyrexia (General disorders) | 130 | 111 | 19 | 5 | 7 | 13 | 91 | 2 | 17
Nasopharyngitis (Infections and infestations) | 50 | 49 | 1 | 6 | 3 | 6 | 29 | 2 | 10
Alanine aminotransferase increased (Investigations) | 101 | 91 | 10 | 9 | 4 | 20 | 69 | 1 | 7
Amylase increased (Investigations) | 39 | 35 | 4 | 2 | 1 | 5 | 29 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 85 | 77 | 8 | 8 | 4 | 16 | 59 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 28 | 26 | 2 | 3 | 3 | 6 | 18 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 28 | 26 | 2 | 5 | 1 | 1 | 24 | 1 | 1
Lipase increased (Investigations) | 75 | 68 | 7 | 10 | 4 | 6 | 57 | 0 | 8
Weight decreased (Investigations) | 53 | 49 | 4 | 3 | 4 | 4 | 41 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 115 | 108 | 7 | 12 | 7 | 10 | 85 | 1 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 40 | 36 | 4 | 5 | 2 | 7 | 27 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 75 | 73 | 2 | 5 | 2 | 9 | 52 | 1 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 49 | 45 | 4 | 6 | 1 | 3 | 40 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 29 | 28 | 1 | 2 | 1 | 3 | 20 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 36 | 4 | 2 | 2 | 4 | 28 | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 | 33 | 3 | 2 | 6 | 4 | 19 | 3 | 4
Headache (Nervous system disorders) | 117 | 110 | 7 | 13 | 5 | 13 | 87 | 3 | 9
Insomnia (Psychiatric disorders) | 58 | 52 | 6 | 5 | 3 | 4 | 47 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 108 | 98 | 10 | 7 | 3 | 12 | 78 | 2 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 59 | 56 | 3 | 3 | 4 | 5 | 40 | 2 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 146 | 135 | 11 | 11 | 11 | 13 | 102 | 4 | 16
Rash (Skin and subcutaneous tissue disorders) | 82 | 76 | 6 | 5 | 4 | 7 | 59 | 3 | 9
Rash macular (Skin and subcutaneous tissue disorders) | 33 | 31 | 2 | 2 | 4 | 2 | 23 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 64 | 58 | 6 | 5 | 3 | 5 | 49 | 2 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 33 | 31 | 2 | 0 | 3 | 1 | 28 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 67 | 58 | 9 | 7 | 2 | 1 | 54 | 1 | 9
Hypertension (Vascular disorders) | 27 | 27 | 0 | 1 | 1 | 6 | 17 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT02599402/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT02599402/SAP_001.pdf